CLINICAL TRIAL: NCT00363142
Title: See Detailed Description.
Brief Title: A Study of an Investigational Regimen Combining FDA Approved HIV Drugs in HIV-Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEX106430
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection; Infection, Human Immunodeficiency Virus
Keywords: HIV-1 LEXIVA Ritonavir Once-daily
MeSH Terms: conditions — HIV Infections; Infections; Acquired Immunodeficiency Syndrome | interventions — fosamprenavir; Ritonavir

ARMS (2):
- FPV/r200 (Active Comparator): Fosamprenavir/ritonavir (either 700/100mg BID or 1400/200mg QD)
  Interventions: Drug: Full Boosted Fosamprenavir
- FPV/r100 (Experimental): Fosamprenavir/ritonavir 1400/100mg QD
  Interventions: Drug: Half-boosted Fosamprenavir

INTERVENTIONS:
Drug: Half-boosted Fosamprenavir — Once daily, reduced dose ritonavir-boosted fosamprenavir
  Arms: FPV/r100
Drug: Full Boosted Fosamprenavir — Full ritonavir-boosted fosamprenavir
  Other Names: Fosamprenavir; ritonavir
  Arms: FPV/r200

SUMMARY:
This is a 24-week study to evaluate the efficacy and safety of a once-daily ritonavir-boosted fosamprenavir regimen (1400mg/100mg QD) to a 200mg ritonavir-boosted fosamprenavir regimen administered either twice-daily or once-daily.

DETAILED DESCRIPTION:
A Phase IIIB, randomized, open-label, parallel group, multi-center, non-inferiority, 24-week study to evaluate the safety, efficacy and tolerability of switching from a 200mg ritonavir-boosted regimen of LEXIVA (700mg/100mg BID or 1400mg/200mg QD) to a once-daily, 100mg ritonavir-boosted regimen of LEXIVA (1400mg/100mg QD)

ELIGIBILITY:
Inclusion criteria:

* Subjects with HIV-1 infection.
* Are willing and able to understand and provide written consent prior to participation in this study.

Exclusion criteria:

* Are pregnant or breastfeeding.
* Have an active AIDS condition, pancreatitis, poor kidney function, or clinically relevant hepatitis.
* Have certain medical conditions that may make participation unsafe.
* Take medication that may interact with the study medication.
* Have a history of allergy to any of the study drugs or any excipients therein.
* Other inclusion/exclusion criteria to be evaluated by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United States (42):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, West Hollywood, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Harlingen, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Spokane, Washington
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan

REFERENCES:
- [Derived] Cohen C, Dejesus E, Lamarca A, Young B, Yau L, Patel L, Vavro C, Wire MB, Wannamaker P, Shaefer M. Similar virologic and immunologic efficacy with fosamprenavir boosted with 100 mg or 200 mg of ritonavir in HIV-infected patients: results of the LESS trial. HIV Clin Trials. 2010 Sep-Oct;11(5):239-47. doi: 10.1310/hct1105-239. PMID 21126954

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified prior to randomization according to baseline regimen (700 milligrams [mg]/100 mg twice a day [BID] or 1400 mg/200 mg once a day [QD]) and previous regimen (no other prior protease inhibitor [PI], non-boosted PI, or boosted PI). Results are reported for the 209 participants (out of 211 enrolled) receiving study drug.
Groups:
- FPV/r100: Fosamprenavir (FPV)/ritonavir (RTV) 1400mg/100mg once a day (QD)
- FPV/r200: FPV/RTV (either 700mg/100mg twice a day [BID] or 1400mg/200mg QD)
Period: Overall Study
Arm/Group | FPV/r100 | FPV/r200
Started | 140 | 69
Completed | 133 | 66
Not Completed | 7 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FPV/r100 | FPV/r200 | Total
Number analyzed (Participants) | 140 | 69 | 209
Age Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.52) | 44.3 (8.9) | 44.7 (10.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 9 | 42
  Male | 107 | 60 | 167
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African heritage | 42 | 20 | 62
  American Indian/Alaskan native | 1 | 0 | 1
  Asian - South East Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White - Arabic/North African | 0 | 2 | 2
  White - White/Caucasian/European | 95 | 44 | 139
  Mixed race | 1 | 0 | 1
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 11 | 42
  Not Hispanic or Latino | 109 | 58 | 167
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Not Meeting the Definition of Virologic Failure at or Prior to Week 24
Description: Virologic failure was defined as two consecutive plasma HIV-1 RNA measures greater than 400 copies/milliliter (mL) separated by at least 2 to 4 week. The percentage of participants not meeting the virologic failure definition was estimated with stratification by the six randomization strata using Mantel-Haenszel weights and the missing/discontinuation equals failure (MD=F) analysis. Missing/discontinuation values were considered failures.
Time Frame: Week 24
Population: Intent-to-Treat Exposed (ITT-E) Population. Subjects who received at least one dose of investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 140 | 69
Percentage of participants | 92.1 | 94.2
Statistical Analysis 1: Comparison: FPV/r100 vs FPV/r200; Test type: Non-Inferiority or Equivalence — Non-inferiority of FPV/r100 to FPV/r200 would be declared if the lower limit of the 2-sided 95% confidence interval on the difference in percentage of participants not meeting the virologic failure definition [FPV/r100 minus FPV/r200] was -12% or greater; Difference in the percentages = -2.12, 95% CI [-9.36 to 5.12] — Difference in percentages = percentage in Arm 1 minus percentage in Arm 2

2. Secondary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus, Type 1, Ribonucleic Acid (HIV-1 RNA) <400 Copies/mL at Week 24, Time to Loss of Virologic Response (TLOVR) Analysis
Description: A blood sample was drawn to determine the amount of plasma HIV-1 RNA virus in copies/mL at week 24. The percentage of participants with plasma HIV-1 RNA <400 copies/mL at Week 24 were determined by the TLOVR algorithm with stratification by the six randomization strata.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 140 | 69
Percentage of participants
  Plasma HIV-1 RNA <400 copies/mL | 92 | 94.2
  HIV-1 RNA greater than or equal to 400 copies/mL | 8 | 5.8

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL at Week 24, TLOVR Analysis
Description: A blood sample was drawn to determine the amount of plasma HIV-1 RNA virus in copies/mL at week 24. The percentage of participants plasma with HIV-1 RNA <50 copies/mL at Week 24 were determined by the TLOVR algorithm with stratification by the six randomization strata.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 140 | 69
Percentage of participants
  Plasma HIV-1 RNA <50 copies/mL | 82.9 | 84.6
  HIV-1 RNA greater than or equal to 50 copies/mL | 17.1 | 15.4

4. Secondary Outcome: Mean Change From Baseline of log10 Copies/mL Plasma HIV-1 RNA Levels at Week 24, Observed Analysis
Description: A blood sample was drawn to determine the amount of plasma HIV-1 RNA virus in copies/mL at week 24. Change from baseline was defined as plasma HIV-1 RNA level at Week 24 minus plasma HIV-1 RNA level at baseline.
Time Frame: Baseline and Week 24
Population: ITT-E Population - Observed Analysis, available data from those subjects who had values at baseline and at Week 24
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 131 | 66
log10 copies/mL | -0.015 (0.388) | -0.022 (0.130)

5. Secondary Outcome: Median Change From Baseline of CD4+ Cell Count at Week 24, Observed Analysis
Description: A blood sample was drawn to determine the CD4+ cell count at week 24. Change from baseline was defined as CD4+ cell count at Week 24 minus CD4+ cell count at baseline.
Time Frame: Baseline and Week 24
Population: ITT-E Population - Observed Analysis, available data from those subjects who had values at baseline and at Week 24
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 132 | 67
cells/mm3 | 11.5 (0.073) [-386 to 407] | 15 (0.194) [-201 to 454]

6. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to Adverse Events Through Week 24
Description: The number of participants who prematurely discontinued study drug due to adverse events was tabulated. Data are summarized by individual adverse event. Adverse events were defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline through Week 24
Population: Safety Population: all randomized subjects who consumed at least one dose of study drug and was analyzed according to the treatment received.
Measure: Number; unit: participants
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 142 | 67
participants
  Any event | 2 | 0
  Alanine aminotransferase increased | 1 | 0
  Aspartate aminotransferase increased | 1 | 0
  Metastatic neoplasms | 1 | 0
  Central nervous system lesion | 1 | 0

7. Secondary Outcome: Number of Participants With Grade 2-4 Adverse Events Occurring in Greater Than or Equal to 2% of Subjects Through Week 24
Description: The number of participants who experienced any grades 2 to 4 adverse events was tabulated. Adverse events were graded based on the Division of Acquired Immunodeficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events.
Time Frame: Baseline through Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 142 | 67
participants
  Any event | 48 | 24
  Diarrhea | 8 | 2
  Bronchitis | 3 | 3
  Nausea | 3 | 1
  Sinusitis | 3 | 1
  Upper respiratory tract infection | 4 | 0
  Blood glucose increased | 3 | 0
  Depression | 1 | 2
  Headache | 1 | 2
  Influenza | 1 | 2
  Low density lipoprotein increased | 3 | 0
  Nasopharyngitis | 3 | 0
  Otitis media | 1 | 2
  Back pain | 0 | 2
  Hypercholesterolemia | 0 | 2
  Insomnia | 0 | 2

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol, High Density Lipoprotein (HDL), and Triglycerides at Week 24
Description: A blood sample was drawn to determine the cholesterol, HDL, triglycerides levels at Week 24. Percent change in total blood cholesterol, HDL, and triglycerides was defined as (lipid level at Week 24 minus level at baseline) divided by level at baseline x 100%.
Time Frame: Baseline and Week 24
Population: Safety Population
Measure: Median (Full Range); unit: Percent change
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 123 | 60
Percent change
  Total cholesterol | -0.5 [-41.8 to 31.3] | 0.7 [-35.4 to 91]
  HDL | -2.1 [-34.8 to 47.4] | 0 [-34.1 to 31.7]
  Triglycerides | -13.5 [-87.7 to 169.2] | -0.6 [-52.2 to 191.1]

9. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein (LDL) at Week 24
Description: A blood sample was drawn to determine the LDL level at Week 24. Percent change in LDL was defined as (LDL level at Week 24 minus level at baseline) divided by level at baseline x 100%.
Time Frame: Baseline and Week 24
Population: Safety Population
Measure: Median (Full Range); unit: Percent change
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 115 | 56
Percent change | 0 [-47 to 103.8] | 2.1 [-60.5 to 142.2]

10. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA Genotypic Mutations and Phenotypic Resistance at Time of Virologic Failure Not Present at Baseline
Description: A blood sample was drawn for subjects failing to respond to therapy and the mutations present in the virus were identified. For each subject, the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New mutations that developed at the time of virologic failure were tabulated by drug class.
Time Frame: Baseline through Week 24
Population: Participants in the ITT-E Population who met the virologic failure definition
Measure: Number; unit: Participants
Arm/Group | FPV/r100 | FPV/r200
Number analyzed (Participants) | 0 | 1
Participants |  | 0

11. Secondary Outcome: Steady-State Plasma Levels of Amprenavir (APV) and Ritonavir (RTV) Ctau at Weeks 12 and 24
Description: Blood samples were drawn at weeks 12 and 24 to determine the plasma levels of APV and RTV. Concentration at the end of the dosing interval at steady state (Ctau) was presented.
Time Frame: Weeks 12 and 24
Population: PK Parameter (Ctau) Population - Participants in the ITT-E Population who underwent PK sampling and had evaluable APV or RTV Ctau data.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Groups:
- FPV/r100: Fosamprenavir (FPV)/ritonavir (RTV) 1400/100mg once a day (QD)
- FPV/r200: FPV/RTV (either 700/100mg twice a day [BID] or 1400/200mg QD)
- FPV/RTV 700/100 mg BID: Twice daily FPV regimen boosted with a reduced dose of RTV 100 mg
Arm/Group | FPV/r100 | FPV/r200 | FPV/RTV 700/100 mg BID
Number analyzed (Participants) | 61 | 17 | 17
micrograms/mL
  Week 12 APV Ctau | 1.38 [1.09 to 1.74] | 1.28 [0.69 to 2.37] | 1.35 [0.44 to 4.11]
  Week 24 APV Ctau | 1.27 [0.99 to 1.62] | 1.49 [1.02 to 2.18] | 2.38 [1.68 to 3.37]
  Week 12 RTV Ctau | 0.026 [0 to 0.286] | 0.050 [0 to 0.346] | 0.228 [0 to 0.568]
  Week 24 RTV Ctau | 0.022 [0 to 2.49] | 0.056 [0 to 0.634] | 0.203 [0 to 1.10]

ADVERSE EVENTS:
Arm/Group | FPV/r100 | FPV/r200
Serious Adverse Events (participants affected / at risk) | 7 | 1
Other Adverse Events (participants affected / at risk) | 18 | 6
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | FPV/r100 | FPV/r200
Pancreatitis chronic (Gastrointestinal disorders) | 1/142 | 0/67
Peptic ulcer (Gastrointestinal disorders) | 1/142 | 0/67
Appendicitis (Infections and infestations) | 1/142 | 0/67
Cellulitis (Infections and infestations) | 1/142 | 0/67
Central nervous system lesion (Nervous system disorders) | 1/142 | 0/67
Cerebrovascular accident (Nervous system disorders) | 1/142 | 0/67
Cardiac failure congestive (Cardiac disorders) | 1/142 | 0/67
Chest pain (General disorders) | 0/142 | 1/67
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/142 | 0/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | FPV/r100 | FPV/r200
Diarrhea (Gastrointestinal disorders) | 9/142 | 4/67
Upper respiratory tract infection (Infections and infestations) | 10/142 | 2/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.